CLINICAL TRIAL: NCT00586495
Title: Extension Study for BAY43-9006 in Japanese Patients With Renal Cell Carcinoma
Brief Title: Long-term Extension From RCC Phase II (11515)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12056
Record Dates: First submitted 2007-12-21; First posted 2008-01-04 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Sorafenib; Nexavar; Metastatic RCC; Renal Cell Carcinoma; Unresectable RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sorafenib (Nexavar, BAY43-9006) (Experimental): Sorafenib 200 mg tablets (400 mg [2 x 200 mg tablets] twice daily [bid] or 400 mg once daily [od] or 400 mg every other day [qod]) administered orally
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Sorafenib 200 mg tablets (400 mg [2 x 200 mg tablets] twice daily [bid] or 400 mg once daily [od] or 400 mg every other day [qod]) administered orally

SUMMARY:
Extension to study 11515 (NCT00661375) which was a multicenter study of sorafenib in patients with renal cell carcinoma (RCC).

ELIGIBILITY:
Inclusion Criteria:

Patients are classified into two groups as below at transition date from Study 11515 to this study.

Population I: Patients who are willing to continue the study drug, for whom the investigator consider continuation of the study drug is appropriate, and who do not meet the criteria of removal from the study in Study 11515 at the end of Study 11515.

Population II: Patients who have been monitored only for survival status at the end of Study 11515.

Population 1

1. Patients who are willing to continue the study drug,
2. Patients for whom the investigator consider continuation of the study drug is appropriate
3. Patients who do not meet the criteria of removal from the study in Study 11515 at the end of Study 11515.
4. Patients who give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Population 2

1. Patients who give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.

Exclusion Criteria:

1. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
2. Any condition that could jeopardize the safety of the patient or that affect his/her compliance in the study
3. Pregnant or breast-feeding patients. Both men and women enrolled in this trial must use adequate birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2005-12; Primary Completion 2008-06 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (36):
- Japan (36):
  - Akita, Akita
  - Asahi, Chiba
  - Chiba, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kurume, Fukuoka
  - Isesaki, Gunma
  - Maebashi, Gunma
  - Sapporo, Hokkaido
  - Sunagawa, Hokkaido
  - Tsukuba, Ibaraki
  - Morioka, Iwate
  - Kagoshima, Kagoshima-ken
  - Kyoto, Kyoto
  - Tsu, Mie-ken
  - Natori-shi, Miyagi
  - Kashihara, Nara
  - Kurashiki, Okayama-ken
  - Okayama, Okayama-ken
  - Osaka, Osaka
  - Sayama, Osaka
  - Suita, Osaka
  - Hidaka, Saitama
  - Irima-gun, Saitama
  - Tokorozawa, Saitama
  - Hamamatsu, Shizuoka
  - Sunto, Shizuoka
  - Utsunomiya, Tochigi
  - Tokushima, Tokushima
  - Arakawa-ku, Tokyo
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Yamagata, Yamagata
  - Ube, Yamaguchi

REFERENCES:
- [Result] Naito S, Tsukamoto T, Murai M, Fukino K, Akaza H. Overall survival and good tolerability of long-term use of sorafenib after cytokine treatment: final results of a phase II trial of sorafenib in Japanese patients with metastatic renal cell carcinoma. BJU Int. 2011 Dec;108(11):1813-9. doi: 10.1111/j.1464-410X.2011.10281.x. Epub 2011 Apr 11. PMID 21481133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was an extension study of Study 11515 (NCT00661375), in which the first subject was enrolled on 10 Nov 2004. This extension study was started in December 2005, and the last subject completed the study on 11 Jul 2008. The study was conducted in 41 centers in Japan.
Pre-assignment Details: 95 subjects were enrolled in this extension study; 95 were valid for the safety analysis and 94 were valid for the intent-to treat (ITT) analysis. 92 subjects entered Follow-up period which started 30 days after last dose. 3 subjects did not enter the Follow-up period because they died within 30 days after last dose.
Period: Treatment Period
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 95
Completed | 0
Not Completed | 95
Not completed — Adverse Event | 11
Not completed — Death | 1
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1
Not completed — Disease progression, recurrence/relapse | 71
Not completed — Switch to commercial drug | 10
Period: Follow-up
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Started | 92
Completed | 0
Not Completed | 92
Not completed — Death | 40
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Protocol driven decision point | 37
Not completed — Switch to commercial drug | 10

BASELINE CHARACTERISTICS:
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 95
Age Continuous [Mean (Standard Deviation); unit: years] | 62.0 (10.5)
Age, Customized [Number; unit: participants]
  <65 years | 54
  >=65 years | 41
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 74
Eastern Cooperative Oncology Group (ECOG) performance status [Number; unit: participants] — ECOG performance status is a rating of daily living abilities, from 0 to 5. 0=Fully active without restriction. 1= Restricted in physically strenuous activity. 2= Ambulatory, capable of all selfcare. 3=Capable of limited selfcare. 4= Completely disabled. 5= Dead.
  participants
    0 | 80
    1 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time from initiation of treatment to disease progression (radiological or clinical, whichever earlier) or death (if death occurs before progression).
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 8 weeks
Population: Intention to treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
days | 386 [274 to 502]

2. Secondary Outcome: Best Tumor Response
Description: Best tumor response, including Complete Response (CR: Disappearance of all target lesions) or Partial Response (PR: At least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum longest diameter) according to the Response Evaluation Criteria in Solid Tumors (RECIST)
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 8 weeks
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
participants
  Complete Response (CR) | 0
  Partial Response (PR) | 25
  Stable Disease (SD) | 64
  Disease Progression (radiological or clinical) | 4
  Not evaluated | 1

3. Secondary Outcome: Overall Survival (OS)
Description: Time from initiation of treatment to death due to any cause.
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 3 months
Population: ITT population. The median overall survival (OS) and the lower limit of 95% Confidence interval were not estimable because more than half (n=51) of the study population were censored. The number of participant who died is shown in "Post-Hoc Outcome Measure: Number of Participants who Died".
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Duration
Description: Time from the date of first objective response (CR or PR, whichever is first recorded) to the date when progressive disease (PD, at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions) is first documented according to RECIST.
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 8 weeks
Population: ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
days | 419 [238 to 862]

5. Secondary Outcome: Time to Objective Response
Description: Time from initiation of treatment to the date when an objective response (CR or PR, whichever is first recorded) is first documented according to RECIST.
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 8 weeks
Population: ITT population.
Measure: Median (Full Range); unit: days
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
days | 84 [35 to 558]

6. Secondary Outcome: Overall Disease Control
Description: Subjects who have a best response rating of CR, PR or Stable Disease (SD: Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum longest diameter since the treatment started) per RECIST that is maintained for at least 28 days from the first demonstration of that rating.
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 8 weeks
Population: ITT population.
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
participants | 81

7. Post Hoc Outcome: Number of Participants Who Died
Description: Number of subjects who died due to any cause.
Time Frame: From start of treatment of the first subject until 45 months later, assessed every 3 months
Population: "Overall Survival" is shown in "Secondary Outcome Measure: Overall Survival".
Measure: Number; unit: participants
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Number analyzed (Participants) | 94
participants | 43

ADVERSE EVENTS:
Description: Acronyms used in Adverse Event section: Absolute Neutrophil Count (ANC), Alanine Transaminase (ALT), Aspartate Transaminase (AST), Common Terminology Criteria for Adverse Events (CTCAE), Creatine Phosphokinase (CPK), Gamma-Glutamyl Transpeptidase (GGT), Gastro-Intestinal (GI), Not Otherwise Specified (NOS).
Arm/Group | Sorafenib (Nexavar, BAY43-9006)
Serious Adverse Events (participants affected / at risk) | 34/95
Other Adverse Events (participants affected / at risk) | 95/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=95)
Hemoglobin (Blood and lymphatic system disorders) | 2
Leukocytes (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 1
Prolonged QTC (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 2
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Constitutional symptoms - other (General disorders) | 1
Fever (General disorders) | 1
Death not associated with CTCAE term, death NOS (General disorders) | 1
Death not associated with CTCAE term, disease progression NOS (General disorders) | 1
Anorexia (Gastrointestinal disorders) | 3
Dehydration (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Distension (Gastrointestinal disorders) | 1
GI - other (Gastrointestinal disorders) | 2
Ileus (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Ulcer, GI, duodeum (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hemorrhage pulmonary, bronchus (Vascular disorders) | 1
Hemorrhage, GI, colon (Vascular disorders) | 1
Hemorrhage, GI, duodenum (Vascular disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Liver dysfunction (Hepatobiliary disorders) | 2
Infection - other (Infections and infestations) | 1
Infection with normal ANC, bronchus (Infections and infestations) | 1
Infection with normal ANC, lung (pneumonia) (Infections and infestations) | 3
Infection with normal ANC, upper airway NOS (Infections and infestations) | 1
Edema: limb (Blood and lymphatic system disorders) | 2
Lymphatics - other (Blood and lymphatic system disorders) | 1
ALT (Metabolism and nutrition disorders) | 2
Amylase (Metabolism and nutrition disorders) | 1
AST (Metabolism and nutrition disorders) | 2
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 1
CPK (Metabolism and nutrition disorders) | 1
GGT (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Lipase (Metabolism and nutrition disorders) | 2
Metabolic/lab - other (Metabolism and nutrition disorders) | 2
Proteinuria (Metabolism and nutrition disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Cataract (Eye disorders) | 1
No code in CTCAE (General disorders) | 3
Pain, abdomen NOS (General disorders) | 1
Pain, tumor pain (General disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1
Syndromes - other (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sorafenib (Nexavar, BAY43-9006) (N=95)
Allergic reaction (Immune system disorders) | 6
Auditory/ear - other (Ear and labyrinth disorders) | 5
Blood - other (Blood and lymphatic system disorders) | 5
Hemoglobin (Blood and lymphatic system disorders) | 14
Leukocytes (Blood and lymphatic system disorders) | 7
Lymphopenia (Blood and lymphatic system disorders) | 8
Hypertension (Cardiac disorders) | 41
Fatigue (General disorders) | 31
Fever (General disorders) | 19
Hypothermia (General disorders) | 7
Insomnia (General disorders) | 8
Rigors/chills (General disorders) | 6
Weight loss (General disorders) | 28
Alopecia (Skin and subcutaneous tissue disorders) | 48
Dermatology - other (Skin and subcutaneous tissue disorders) | 15
Dry skin (Skin and subcutaneous tissue disorders) | 6
Flushing (Skin and subcutaneous tissue disorders) | 5
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 61
Pruritus (Skin and subcutaneous tissue disorders) | 19
Rash/desquamation (Skin and subcutaneous tissue disorders) | 54
Hot flashes (Endocrine disorders) | 5
Anorexia (Gastrointestinal disorders) | 27
Constipation (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 58
Distension (Gastrointestinal disorders) | 5
GI - other (Gastrointestinal disorders) | 5
Heartburn (Gastrointestinal disorders) | 9
Mucositis (clinical exam), oral cavity (Gastrointestinal disorders) | 6
Mucositis (functional/symptomatic), oral cavity (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 15
Periodontal (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 16
Hemorrhage pulmonary, bronchopulmonary NOS (Vascular disorders) | 6
Hemorrhage pulmonary, nose (Vascular disorders) | 7
Infection - other (Infections and infestations) | 12
Infection with normal ANC, Bronchus (Infections and infestations) | 5
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 12
Edema: head and neck (Blood and lymphatic system disorders) | 7
Edema: limb (Blood and lymphatic system disorders) | 16
Alkaline phosphatase (Metabolism and nutrition disorders) | 15
ALT (Metabolism and nutrition disorders) | 23
Amylase (Metabolism and nutrition disorders) | 43
AST (Metabolism and nutrition disorders) | 24
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 5
Creatinine (Metabolism and nutrition disorders) | 8
GGT (Metabolism and nutrition disorders) | 7
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 11
Lipase (Metabolism and nutrition disorders) | 62
Metabolic/lab - other (Metabolism and nutrition disorders) | 38
Proteinuria (Metabolism and nutrition disorders) | 12
Musculoskeletal - other (Musculoskeletal and connective tissue disorders) | 12
Dizziness (Nervous system disorders) | 6
Neuropathy - sensory (Nervous system disorders) | 6
Ocular surface disease (Eye disorders) | 5
Pain, abdomen NOS (General disorders) | 11
Pain, back (General disorders) | 23
Pain, chest/thorax NOS (General disorders) | 10
Pain, dental/teeth/peridontal (General disorders) | 5
Pain, extremity/limb (General disorders) | 13
Pain, head/headache (General disorders) | 18
Pain, joint (General disorders) | 16
Pain, other (General disorders) | 8
Pain, stomach (General disorders) | 6
Pain, throat/pharynx/larynx (General disorders) | 10
Pain, tumor pain (General disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 21
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 5
Voice changes (Respiratory, thoracic and mediastinal disorders) | 18
Flu-like syndrome (General disorders) | 34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less